CLINICAL TRIAL: NCT02261519
Title: An Adaptive, Phase IIb/III, Multi-center, Prospective, Randomized, Double-Blind Placebo-controlled Study of the Safety and Efficacy of NaBen® (DAAO Inhibitor), as an Add-on Treatment for Schizophrenia in Adults
Brief Title: Study to Evaluate Safety & Efficacy of NaBen® as Add-on Treatment for Schizophrenia in Adults
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: due to commercial strategy
Sponsor: SyneuRx International (Taiwan) Corp (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SNR-04
Record Dates: First submitted 2014-09-25; First posted 2014-10-10 (Estimated); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NaBen® (Experimental): NaBen® is a oral tablet (500 mg), which will be taken twice daily at a total dose of 1000 mg/day during this study.
  Interventions: Drug: NaBen®
- Placebo (Placebo Comparator): The control treatment is placebo.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: NaBen® — 500 mg twice daily (1000 mg total)
  Arms: NaBen®
Other: Placebo — 0 mg twice daily (0 mg total)
  Arms: Placebo

SUMMARY:
The proposed Phase IIb/III study is designed to evaluate the safety and efficacy of NaBen® in improving the symptoms of schizophrenia in adults. NaBen® is granted Breakthrough Therapy Designation by US FDA as add-on treatment for schizophrenia. The trial is designed as a multi-center, prospective, randomized, placebo-controlled, in which adult subjects with schizophrenia will be enrolled. The study will include four parts: a 2 week Screening part, a 4 week run-in part, an 8 week double-blind treatment part, and a 52 week Open-Label Extension part.

DETAILED DESCRIPTION:
This is an adaptive, phase IIb/III, multi-center, prospective, randomized, placebo-controlled study, in which adult subjects with schizophrenia will be enrolled. The study will include four parts: a 2 week Screening part, a 4 week run-in part, and 8 week double-blind treatment part, and a 52 week Open-Label Extension part.

Screening part of the study:

The subjects will be evaluated for eligibility during the Screening part of the study.

Enrichment run-in part of the study:

Subjects who are determined to be eligible will enter the Run-in part of the study. A total of 348 Subjects will be randomized. The randomized subjects will receive 4 weeks of NaBen® or Placebo accordingly. The subjects who have completed 4 weeks of randomized treatment in both groups (NaBen® or Placebo) will be assessed and categorized intoresponders and non-responders, based on 20% or more reduction from baseline in their PANSS total scores as per the evaluations at Visit 2 and Visit 4.

Double-Blind treatment part of the study :

* Subjects who have successfully completed the Enrichment Run-in part will enter the Double- Blind treatment part of the study per below: NaBen® treated subjects: Subjects will continue receiving NaBen® for another 8 weeks.
* Placebo treated subjects:

  * Placebo Responders: Subjects will continue receiving Placebo for another 8 weeks.
  * Placebo Non-responders: Subjects will be re-randomized to receive NaBen® or Placebo in a 1:1 ratio for another 8 weeks.

Open-Label Extension part of the study:

All subjects who have completed the Double-Blind part of the study will continue with the Open-Label Extension part of the study to receive NaBen® for an additional 52 weeks, plus a 2 week follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Male/female subjects between 18 and 45 years of age
2. If female and not infertile (defined below), the subject must agree for the duration of the study to use one of the following forms of contraception 1) systemic hormonal treatment 2) an Intrauterine device (IUD) which was implanted at least 2 months prior to screening or 3) "double-barrier" contraception (condom, diaphragm and spermicide are each considered a barrier). Females are considered to be infertile if they are either a) surgically sterile or b) have had spontaneous amenorrhea for at least the last 2 years and at least 2 years after the onset of amenorrhea while not receiving hormone replacement therapy and had a Follicle-Stimulating Hormone (FSH) level greater than 40 mIU/mL and an estradiol level less than 30 pg/mL
3. Subject is capable of providing informed consent and is willing to sign the ICF prior to study Screening and agrees to comply with the study protocol requirements
4. Physician confirmed DSM-V diagnosis of schizophrenia for the past 2 years based on subject's history and confirmed by psychiatric evaluation and MINI International Neuropsychiatric Interview For Schizophrenia and Psychotic Disorders, version 7.0 (MINI, Version 7.0)
5. The subject is outpatient with no hospitalization for worsening of schizophrenia within 3 months of the screening.If the subject is hospitalized during the study for worsening of schizophrenia symptoms the subject will be withdrawn from the study
6. The subject's schizophrenia condition is clinically stable with residual symptoms. Residual symptoms will be defined as a total score of ≤110 and ≥ 60 of PANSS per Visit 1 evaluations
7. An unchanged antipsychotic medication regimen for at least eight (8) weeks prior to screening into the study and expected to remain unchanged during the study (longer for depot or long-acting antipsychotics: ten (10) months for Aripiprazole and Paliperidone; six (6) months for Olanzapine pamoate monohydrate; and at least 6 times duration of the reported half life or minimum four (4) months for other depot or long-acting antipsychotics)
8. In good general physical health and without clinically significant abnormalities in physical exam, neurological exam and laboratory assessments (urine/blood routine, biochemical tests and ECG) which would exclude the subject from the study in the opinion of the Investigator. For ALT and AST, clinically significant is defined as above twice the upper limit of normal.
9. BMI between 17 and 35 inclusive
10. Subject has a negative routine urine illicit drug screening test (including heroin, amphetamines (including MDMA/ecstasy), cocaine, cannabis or PCP)
11. The subject has a caregiver or some other identified responsible person (e.g., family member, social worker, caseworker or nurse) as determined by the Investigator and per the local regulations. The identified caregiver should be considered reliable by the Investigator and per the local regulations in providing support to the subject to help ensure compliance with study treatment, study visits and protocol procedures who preferably is also able to provide input helpful for completing study rating scales
12. The subject must not be a danger to self or others per the Investigator's judgment

Exclusion Criteria:

1. Meets the DSM-IV or V criteria at screening for intellectual disability, dissociative disorder, bipolar disorder, major depressive disorder, schizoaffective disorder, schizophreniform disorder, autistic disorder, primary substance-induced psychotic disorder, dementia, or any other comorbid mental disorders that in the opinion of the Investigator may interfere with study conduct and results interpretation
2. Subjects whose illness was resistant to antipsychotics according to prior trials of two different antipsychotics of adequate dose
3. Subjects who have been previously treated with or are receiving clozapine
4. Initiation or dose change of lithium, antidepressant or other mood stabilizers within 16 weeks prior to screening
5. Initiation or dose change of benzodiazepines or sleep medications due to worsening of schizophrenia symptoms or medication side effects, or any other psychotropic medications within 4 weeks prior to screening
6. The subject has previously received NaBen®
7. History of epilepsy, major head trauma, or any neurological illness other than Tourette's syndrome which might impair the subject's cognition or psychiatric functioning per the investigator's judgment
8. History of allergic reaction to sodium benzoate
9. Serious medical illnesses such as end-stage renal disease, liver failure or heart failure that, in the opinion of the Investigator, may interfere with the conduct of the study
10. Any significant gastrointestinal disorders that, in the opinion of the investigator, markedly alter the absorption, metabolism or elimination of sodium benzoate
11. Any movement disorders with a total score higher than 6 on SAS scale, or more than 2 on any items of the AIMS scale
12. Current substance abuse, or history of meeting criteria for moderate or severe substance abuse (including alcohol, but excluding nicotine and caffeine) in the past six (6) months prior to screening
13. Female subjects who are pregnant (as confirmed by urine pregnancy test performed at Screening Visit) or are breast feeding
14. History of cancer not in remission for the last 3 years except for basal cell carcinoma and squamous cell carcinoma
15. Participation in a clinical trial within 3 months prior to screening or more than two clinical trials within 12 months
16. Electroconvulsive Therapy within 6 months prior to screening
17. The subject started a new non-medication treatment for schizophrenia or other psychiatric condition within the last 3 months prior to screening
18. The subject's anti-EPS medications dose or regimen has changed within 2 weeks prior to screening

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 280 (Actual)
Dates: Start 2017-03-29 (Actual); Primary Completion 2023-11-29 (Actual); Study Completion 2023-11-29 (Actual)

PRIMARY OUTCOMES:
Positive and Negative Syndrome Scale (PANSS) | 8 weeks after randomized treatment
  Mean change from baseline in PANSS total score

SECONDARY OUTCOMES:
Positive and Negative Syndrome Scale (PANSS) | 8 weeks after treatment
  Percent change from baseline in PANSS total score
Positive and Negative Syndrome Scale (PANSS) | 8 weeks after treatment
  Percentage of subjects with 20% or more reduction from baseline in PANSS total score
PANSS sub-scale scores and Marder PANSS factor scores | 8 weeks after treatment
  Percent change in PANSS sub-scale scores and Marder PANSS factor scores
Personal and Social Performance (PSP) scale | 8 weeks after treatment
  Percent change of Personal and Social Performance (PSP) scale

OTHER OUTCOMES:
Positive and Negative Syndrome Scale (PANSS) | 64 weeks
  Maintenance of treatment effect for PANSS total score
Personal and Social Performance (PSP) scale | 64 weeks
  Maintenance of treatment effect in PSP scale
Schizophrenia Quality of Life Scale (SQLS) | 64 weeks
  Percent change and maintenance of treatment effect in Schizophrenia Quality of Life Scale (SQLS)
Clinical Global Impression-Severity (CGI-S) and -improvement (CGI-I) | 64 weeks
  Percent change and maintenance of treatment effect in Clinical Global Impression-Severity (CGI-S) and -improvement (CGI-I) for both overall and negative symptoms
Hamilton Depression Rating Scale (HDRS) | 64 weeks
  Percent change in Hamilton Depression Rating Scale (HDRS)
Serum analysis | 12 weeks
  Serum pharmacokinetic evaluations, DNA evaluations and neurotransmitter markers evaluations
Treatment-Emergent Adverse Events (TEAE) | 64 weeks
  Incidence of TEAE and incidence of withdrawals from the study due to TEAEs
Simpson-Angus extrapyramidal side effects (SAS) scale | 64 weeks
  Percent change in Simpson-Angus extrapyramidal side effects (SAS) scale
Abnormal Involuntary Movement Scale (AIMS) | 64 weeks
  Percent change in Abnormal Involuntary Movement Scale (AIMS)
Barnes Akathisia Rating Scale (BARS) | 64 weeks
  Percent change in Barnes Akathisia Rating Scale (BARS)
Columbia-Suicide Severity Rating Scale (C-SSRS) | 64 weeks
  Assessment of suicidality per the Columbia-Suicide Severity Rating Scale (C-SSRS)
Laboratory measurements (e.g., Hematology, Biochemistry, Urine analysis) | 64 weeks
  Changes and shifts in laboratory measurements (e.g., Hematology, Biochemistry, Urine analysis) over time
Vital signs (e.g., Body temperature, Heart rate, Respiration rate, Blood pressure) | 64 weeks
  Changes in vital signs (e.g., Body temperature, Heart rate, Respiration rate, Blood pressure) over time
Weight (e.g., BMI in kg/m2) | 64 weeks
  Changes in weight (e.g., BMI in kg/m2)over time
Electrocardiogram (ECG) parameters | 64 weeks
  Changes in Electrocardiogram (ECG) parameters over time

CONTACTS AND LOCATIONS:
Locations (1):
- For additional information regarding investigative sites for this trial, contact SyneuRx International Corp., Pasadena, California, United States